CLINICAL TRIAL: NCT03783065
Title: HVPG-guided Laparoscopic Versus Endoscopic Therapy for Variceal Rebleeding in Portal Hypertension: A Multicenter Randomized Controlled Trial (CHESS1803)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southern Medical University, China (Other); Xingtai People's Hospital (Other); Beijing 302 Hospital (Other); LanZhou University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Hepatic Hemodynamic Lab, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHESS1803
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Portal Hypertension; Variceal Rebleeding
Keywords: Variceal Rebleeding; Hepatic venous pressure gradient; Laparoscopic Therapy; Endoscopic Therapy
MeSH Terms: conditions — Hypertension, Portal | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Procedure: Laparoscopic splenectomy and pericardial devascularization Drug: Propranolol
  Interventions: Drug: Propranolol; Procedure: Laparoscopic splenectomy and pericardial devascularization
- Control group (Active Comparator): Procedure: Endoscopic therapy Drug: Propranolol
  Interventions: Drug: Propranolol; Procedure: Endoscopic therapy

INTERVENTIONS:
Drug: Propranolol — Propranolol was administrated orally while keeping monitoring heart rate and blood pressure daily.
Procedure: Laparoscopic splenectomy and pericardial devascularization — Including splenectomy and pericardial devascularizaion under laparoscopy
  Arms: Experimental group
Procedure: Endoscopic therapy — Either endoscopic variceal ligation (EVL) or cyanoacrylate injection was applied according to the condition of varices
  Arms: Control group

SUMMARY:
The development of portal hypertension is a vital event in the natural progression of cirrhosis and is associated with severe complications including gastroesophageal varices bleeding. Cirrhotic patients with hemorrhagic shock and/or liver failure caused by variceal bleeding face a mortality of 5-20%.

Hepatic venous pressure gradient (HVPG) is the recommended golden standard for portal pressure assessment globally with favorable consistency and repeatability. Reducing the HVPG to levels of 12mmHg or below is associated with protection of variceal hemorrhage. An HVPG> 16mmHg indicates a higher risk of death and HVPG ≥ 20mmHg predicts failure to control bleeding, early rebleeding, and death during acute variceal hemorrhage.

The management of portal hypertension has showed a trend of diversification with the development of medication, endoscopy, radiological intervention and liver transplantation. Although medication and endoscopic therapy have achieved preferable effects and are recommended as standard of care for the prevention of variceal rebleeding, patients with HVPG≥ 16mmHg still have a high risk of treatment failure and a high rate of rebleeding. Recent years, early TIPS is recommended as the first-line therapy for the prevention of rebleeding in cirrhotic patients with HVPG≥ 20mmHg. However, for those with HVPG values between 16 to 20mmHg, there is still lack of strong evidence to demonstrate the best practice for the management.

With the rapid advancement of laparoscopic device and technique, the utility of laparoscopic splenectomy and pericardial devascularization showed less surgical trauma, bleeding and complications while retaining dependable effects compared to traditional open surgery, especially for portal hypertension with hypersplenism. In the study, the investigators aim to conduct a multicenter randomized controlled trial to compare the safety and effectiveness of HVPG-guided (16 to 20mmHg) laparoscopic versus endoscopic therapy for variceal rebleeding in patients with portal hypertension.

DETAILED DESCRIPTION:
The development of portal hypertension is a vital event in the natural progression of cirrhosis and is associated with severe complications including gastroesophageal varices bleeding. Cirrhotic patients with hemorrhagic shock and/or liver failure caused by variceal bleeding face a mortality of 5-20%.

Hepatic venous pressure gradient (HVPG) is the recommended golden standard for portal pressure assessment globally with favorable consistency and repeatability. Reducing the HVPG to levels of 12mmHg or below is associated with protection of variceal hemorrhage. An HVPG> 16mmHg indicates a higher risk of death and HVPG ≥ 20mmHg predicts failure to control bleeding, early rebleeding, and death during acute variceal hemorrhage.

The management of portal hypertension has showed a trend of diversification with the development of medication, endoscopy, radiological intervention and liver transplantation. Although medication and endoscopic therapy have achieved preferable effects and are recommended as standard of care for the prevention of variceal rebleeding, patients with HVPG≥ 16mmHg still have a high risk of treatment failure and a high rate of rebleeding. Recent years, early TIPS is recommended as the first-line therapy for the prevention of rebleeding in cirrhotic patients with HVPG≥ 20mmHg. However, for those with HVPG values between 16 to 20mmHg, there is still lack of strong evidence to demonstrate the best practice for the management.

With the rapid advancement of laparoscopic device and technique, the utility of laparoscopic splenectomy and pericardial devascularization showed less surgical trauma, bleeding and complications while retaining dependable effects compared to traditional open surgery, especially for portal hypertension with hypersplenism. In the study, the investigators aim to conduct a multicenter (Shunde Hospital of Southern Medical University, Xingtai People's Hospital, The Fifth Medical Center of Chinese PLA General Hospital, The First Hospital of Lanzhou University) randomized controlled trial to compare the safety and effectiveness of HVPG-guided (16 to 20mmHg) laparoscopic versus endoscopic therapy for variceal rebleeding in patients with portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and/or pathologically diagnosed cirrhosis with portal hypertension
* History of varicial bleeding without receiving endoscopic treatment
* HVPG values between 16-20 mmHg
* ECOG score ≤ 2 or KPS score ≥ 60 during screening
* Voluntarily participated in the study and able to provide written informed consent, understand and willing to comply with the requirements of the study
* Child-Pugh class A or B

Exclusion Criteria:

* Pregnant or breastfeeding women
* Prior known or suspected malignancy (hepatocellular carcinoma, cholangiocarcinoma etc.)
* Limited coagulation situation (Quick< 50%, PTT> 50 sec, thrombocyte count <50000 / μl or disturbed thrombocyte function)
* Massive ascites
* Child-Pugh class C
* Refuse or inadequate for HVPG measurement
* Other situations whose existence judged inadequate for participation by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2022-10-28 (Estimated)

PRIMARY OUTCOMES:
Variceal rebleeding | 1 year
  The occurrence rate of gastroesophageal varices rebleeding within 1-year follow-up

SECONDARY OUTCOMES:
Overall survival | 1 year
  The number of participants still alive 1 year after the therapy
Hepatocellular carcinoma occurrence | 1 year
  The occurrence rate of hepatocellular carcinoma 1 year after the therapy
Venous thrombosis | 1 year
  The occurrence rate of venous thrombosis upon each follow-up
Quality of life score | 1 year
  The quality of life score measured using the 36-item Short Form Health Survey (SF-36) questionnaire upon each follow-up.
Karnofsky score | 1 year
  The Karnofsky score categorized into low (score 10-40), intermediate (50-70), and high (80-100) upon each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Wang, MD, Principal Investigator — Southern Medical University, China; Changzeng Zuo, MD, Principal Investigator — Xingtai People's Hospital; Xun Li, MD, Principal Investigator — LanZhou University; Xiaolong Qi, MD, Study Chair — Nanfang Hospital, Southern Medical University
Locations (4):
- China (4):
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Shunde Hospital, Southern Medical University, Shunde, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei

IPD SHARING:
Plan to Share IPD: Yes
IPD data including age, gender, height, weight, ethnic, past history (including time of bleeding), dignosis, co-morbidity, medication, labortory test results (including blood routine, blood ammonia, clotting time, liver function and renal function), ultrasonic results (including spleen diameter, portal vein diameter, portal vein velocity, splenic vein velocity, etc.), transient elastography results (including liver and spleen stiffness), esophagogastroduodenoscopy results, Child-pugh score, QOL and KPS scores and time of all outcome events will be shared upon publication of this study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available upon publication of this study for 2 years.
Access Criteria: Access application is approved by principal investigators.

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Cremers I, Ribeiro S. Management of variceal and nonvariceal upper gastrointestinal bleeding in patients with cirrhosis. Therap Adv Gastroenterol. 2014 Sep;7(5):206-16. doi: 10.1177/1756283X14538688. PMID 25177367
- [Background] Garcia-Tsao G, Bosch J. Management of varices and variceal hemorrhage in cirrhosis. N Engl J Med. 2010 Mar 4;362(9):823-32. doi: 10.1056/NEJMra0901512. No abstract available. PMID 20200386
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Bosch J, Abraldes JG, Berzigotti A, Garcia-Pagan JC. The clinical use of HVPG measurements in chronic liver disease. Nat Rev Gastroenterol Hepatol. 2009 Oct;6(10):573-82. doi: 10.1038/nrgastro.2009.149. Epub 2009 Sep 1. PMID 19724251
- [Background] Saad WE. Endovascular management of gastric varices. Clin Liver Dis. 2014 Nov;18(4):829-51. doi: 10.1016/j.cld.2014.07.005. Epub 2014 Oct 16. PMID 25438286
- [Background] de Souza AR, La Mura V, Reverter E, Seijo S, Berzigotti A, Ashkenazi E, Garcia-Pagan JC, Abraldes JG, Bosch J. Patients whose first episode of bleeding occurs while taking a beta-blocker have high long-term risks of rebleeding and death. Clin Gastroenterol Hepatol. 2012 Jun;10(6):670-6; quiz e58. doi: 10.1016/j.cgh.2012.02.011. Epub 2012 Feb 22. PMID 22366180
- [Derived] Shao R, Li Z, Wang J, Qi R, Liu Q, Zhang W, Mao X, Song X, Li L, Liu Y, Zhao X, Liu C, Li X, Zuo C, Wang W, Qi X. Hepatic venous pressure gradient-guided laparoscopic splenectomy and pericardial devascularisation versus endoscopic therapy for secondary prophylaxis for variceal rebleeding in portal hypertension (CHESS1803): study protocol of a multicenter randomised controlled trial in China. BMJ Open. 2020 Jun 23;10(6):e030960. doi: 10.1136/bmjopen-2019-030960. PMID 32580978